CLINICAL TRIAL: NCT04559100
Title: Clinical, Radiological, Lung Function, and Quality of Life Characterization of Patients With Severe/Critical Infection by SARS-COV-2 (COVID-19) Virus, After 6 and 12 Months of Hospital Discharge
Brief Title: Long-term Characterization of Patients With Severe/Critical Infection by COVID-19 Virus
Status: Completed | Type: Observational
Sponsor: Fundacion Clinica Valle del Lili (Other)
Responsible Party: Sponsor
Other Study IDs: 1631 COVID-LFT
Record Dates: First submitted 2020-09-17; First posted 2020-09-22 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-05

CONDITIONS: Covid19
Keywords: covid19; lung function; quality of life
MeSH Terms: conditions — COVID-19 | interventions — X-Rays; Spirometry; Walk Test

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Severe and critical COVID-19 survivors: Radiological alterations assessed by chest radiography and/or thoracic computed tomography Lung function alterations assessed by spirometry, diffusing capacity for carbon monoxide, 6 minute walk.
  Quality of life alterations: saint george respiratory questionnaire
  Interventions: Radiation: chest radiography; Radiation: thoracic computed tomography scan; Diagnostic Test: spirometry; Diagnostic Test: Diffusing capacity of carbon monoxide; Diagnostic Test: 6 minute walk test; Diagnostic Test: saint george respiratory questionnaire

INTERVENTIONS:
Radiation: chest radiography — 6 and 12 months after hospital discharge. If the study is normal at 6 months it will not be repeated at 12 months.
Radiation: thoracic computed tomography scan — 6 and 12 months after hospital discharge, if the patient had a CT scan upon admission to the hospital. If the study is normal at 6 months it will not be repeated at 12 months.
Diagnostic Test: spirometry — 6 and 12 months after hospital discharge. If the study is normal at 6 months it will not be repeated at 12 months.
Diagnostic Test: Diffusing capacity of carbon monoxide — 6 and 12 months after hospital discharge. If the study is normal at 6 months it will not be repeated at 12 months.
Diagnostic Test: 6 minute walk test — 6 and 12 months after hospital discharge. If the study is normal at 6 months it will not be repeated at 12 months.
Diagnostic Test: saint george respiratory questionnaire — 6 and 12 months after hospital discharge.

SUMMARY:
A descriptive study to characterize clinical, radiological, lung function and quality of life alterations in patients who survived a severe or critical disease caused by SARS-COV-2 virus, who were treated in the intensive care unit of a high complexity institution in Cali, Colombia.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 19 years old who had a positive test for SARS-COV-2 virus
* Patients with a severe and critical disease by SARS-COV-2, who were treated at the ICU of Fundación Valle del Lili, and survived
* Patients with chest radiography or CT scan at admission to the hospital

Exclusion Criteria:

* Patients who do not sign informed consent.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a severe or critical disease caused by SARS-COV-2 infection who were treated at the ICU of Fundación Valle del Lili and were alive at 6 months of hospital discharge.
Sampling Method: Non-Probability Sample
Enrollment: 112 (Actual)
Dates: Start 2020-11-15 (Actual); Primary Completion 2021-11-11 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
Lung function | 6 months after hospital discharge
  Spirometry in Liters
Lung function | 12 months after hospital discharge
  Spirometry in Liters
Lung function | 6 months after hospital discharge
  Diffusing capacity of carbon monoxide (% predicted)
Lung function | 12 months after hospital discharge
  Diffusing capacity of carbon monoxide (% predicted)
Lung function | 6 months after hospital discharge
  6 min walk test in Meters
Lung function | 12 months after hospital discharge
  6 min walk test in Meters
Radiological alterations | 6 months after hospital discharge
  Alterations in chest radiography
Radiological alterations | 12 months after hospital discharge
  Alterations in chest radiography
Radiological alterations | 6 months after hospital discharge
  Alterations in thoracic CT scan
Radiological alterations | 12 months after hospital discharge
  Alterations in thoracic CT scan
Quality of life alterations | 6 months after hospital discharge
  Saint George Respiratory questionnaire (from 0 to 100 points, higher levels indicating a major health impairment)
Quality of life alterations | 12 months after hospital discharge
  Saint George Respiratory questionnaire (from 0 to 100 points, higher levels indicating a major health impairment)

CONTACTS AND LOCATIONS:
Overall Officials: Fernandez, Principal Investigator — Fundacion Clinica Valle del Lili
Locations (1):
- Fundacion Valle del Lili, Cali, Valle del Cauca Department, Colombia

IPD SHARING:
Plan to Share IPD: Undecided